CLINICAL TRIAL: NCT05435144
Title: The Effects of Supplementation With ElderCraft® Elderberry Extract: A Randomized, Triple-blind, Placebo Controlled Clinical Trial.
Brief Title: Elderberry for Immune Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Artemis International (Unknown); IPRONA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-07-2400
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Upper Respiratory Tract Infection; COVID-19; Flu; Flu Like Illness; Cold
Keywords: elderberry; anthocyanins
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19; Influenza, Human; Common Cold | interventions — elderberry extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive a 13-week supply of ElderCraft® (European black elderberry extract standardized to 15% anthocyanins). Each capsule contains 300mg of extract; participants will take a total of two capsules each day.
  Interventions: Dietary Supplement: Elderberry
- Placebo Arm (Placebo Comparator): Participants will receive a 13-week supply of inert placebo capsules matched for polysaccharide content. Participants will take a total of two capsules each day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Elderberry — European black elderberry extract
  Other Names: ElderCraft; Sambucus nigra
  Arms: Intervention Arm
Other: Placebo — Inactive placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to confirm and quantify the effects of ElderCraft® elderberry extract on immune health.

DETAILED DESCRIPTION:
This study is a randomized double blind, placebo controlled clinical trial. The purpose is to evaluate the between-groups difference in incidence and duration of upper respiratory events and severity of upper respiratory symptoms while supplementing with ElderCraft® elderberry extract.

After attending an orientation session, participants will provide informed consent and be randomized on a 1:1 basis into an intervention group or a placebo group. Each group will consume two capsules daily for 13 weeks. Each intervention capsule contains 300 mg of European black elderberry extract, standardized to 15% anthocyanins.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures and availability for the duration of the study
* Aged 20-65
* Lives in the United States within driving distance of the research center
* In good general health as evidenced by medical history
* BMI <31
* Ability to take oral supplements and willing to commit to taking 2 capsules a day for 3 months
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the intervention period
* Employed full time in an occupation with direct and prolonged exposure to the public (i.e. teacher, healthcare provider, etc) or regularly engaged in high exposure activities.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Current use of the following pharmaceuticals: immunosuppressants
* Pregnancy, trying to conceive or breastfeeding
* Organ transplant recipient
* Known allergic reactions to elderberries
* Positive COVID-19 test within 180 days of the study period
* COVID vaccine of any type scheduled during the intervention period or the week prior to the start of the study
* Receipt of 4+ COVID-19 vaccines
* Current diagnosis or lifetime history of an autoimmune condition (including but not limited to Lupus, Addisons, Graves, Hypothyroidism, Multiple Sclerosis, or Type 1 Diabetes) OR cancer OR chronic kidney disease OR chronic liver disease OR chronic lung disease (i.e. COPD, pulmonary embolism) OR cystic fibrosis OR severe heart disease (i.e. heart failure, coronary artery disease, cardiomyopathy) OR HIV infection OR immunocompromised status OR sickle cell disease OR tuberculosis
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Existing usage of a polyphenol-based supplement, including but not limited to elderberry, cranberry, bilberry, quercetin, or resveratrol.
* Existing usage of an immune supporting supplement such as echinacea, probiotics, elderberry, or any other dietary supplements marketed as immune support.
* Routine dietary consumption of high levels of polyphenols or anthocyanins as determined by dietary intake questionnaire.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-03-28 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Upper Respiratory Symptomatic Days | 13 weeks
  Total number of days with upper respiratory symptoms during the 90 day intervention. Symptoms are measured using the Franklin Immune Scale, which measures the severity of 50 symptoms. Scores range from 0 (symptom not present) to 5 (symptom is severe), with higher scores indicating greater severity.
Incidence of Upper Respiratory Events | 13 weeks
  Total number of upper respiratory events during the 90 day intervention. An event is classified as a series of continuous days with upper respiratory symptoms.
Duration of Upper Respiratory Events | 13 weeks
  Total number of days per upper respiratory event. An event is classified as a series of continuous days with upper respiratory symptoms.
Symptom Severity | 13 weeks
  Average daily symptom score on the Franklin Immune Scale which measures the severity of 50 symptoms. Scores range from 0 (symptom not present) to 5 (symptom is severe), with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Incidence of COVID-19 | 13 weeks
  Total number of COVID-19 diagnoses during the 90 day period, as confirmed through an at-home laboratory verified diagnostic test.
Duration of COVID-19 | 13 weeks
  Total number of days per COVID-19 infection. An event is classified as a series of continuous days with COVID-19 symptoms and the receipt of a positive COVID-19 test.
Severity of COVID-19 | 13 weeks
  Average daily symptom score on the Franklin Immune Scale which measures the severity of 50 symptoms. Scores range from 0 (symptom not present) to 5 (symptom is severe), with higher scores indicating greater severity.
Incidence of influenza | 13 weeks
  Total number of influenza diagnoses during the 90 day period, as confirmed through an in-office diagnostic test.
Duration of influenza | 13 weeks
  Total number of days per influenza infection. An event is classified as a series of continuous days with flu-like symptoms and the receipt of a positive influenza test.
Severity of influenza | 13 weeks
  Average daily symptom score on the Franklin Immune Scale which measures the severity of 50 symptoms. Scores range from 0 (symptom not present) to 5 (symptom is severe), with higher scores indicating greater severity.
Energy Levels | baseline and 13 weeks
  The Franklin Energy Scale measures energy levels across 7 domains, with higher scores indicating greater energy levels. This produces a total energy score, as well as 7 subscores.
Sleep Quality | baseline and 13 weeks
  The Franklin Sleep Scale measures energy levels across 10 domains, with higher scores indicating greater sleep quality.
Cognitive Wellbeing | baseline and 13 weeks
  The Franklin Cognitive Health Scale measures brain health across 7 domains, with higher scores indicating greater cognitive well-being.
Stress Levels | baseline and 13 weeks
  The Franklin Stress Scale measures stress levels across 7 domains, with higher scores indicating greater stress management.

OTHER OUTCOMES:
Digestive Health | baseline and 13 weeks
  The Franklin Digestive Health Scale measures gastrointestinal health across 4 domains, with higher scores indicating greater gastrointestinal health.
Adverse Events | 13 weeks
  Total number of adverse events during the 13 week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No